CLINICAL TRIAL: NCT04573218
Title: Supplementation of Oil Palm Phenolics to Improve Lipid Profile in Subjects With Minor Hyperlipidaemia (Phase 2 Clinical Trial Study)
Brief Title: Supplementation of Oil Palm Phenolics to Improve Lipid Profile in Subjects With Minor Hyperlipidaemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Isa Naina Mohamed (Other)
Collaborators: Malaysia Palm Oil Board (Other Government)
Responsible Party: Sponsor-Investigator, Isa Naina Mohamed, Associate Professor, National University of Malaysia
Organization: National University of Malaysia (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SAPPHIRE
Record Dates: First submitted 2020-09-28; First posted 2020-10-05 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Hyperlipidemias; Hypercholesterolemia
Keywords: oil palm phenolics; lipid profile
MeSH Terms: conditions — Hyperlipidemias; Hypercholesterolemia | interventions — 4-(2-oxapentadeca-4-yne)phenylpropanoic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Placebo Comparator): Glucose.
  Interventions: Drug: Placebo
- Group B (Active Comparator): 250 mg Oil Palm Phenolics.
  Interventions: Dietary Supplement: 250 mg OPP

INTERVENTIONS:
Drug: Placebo — The placebo contains glucose
  Arms: Group A
Dietary Supplement: 250 mg OPP — 250 mg Oil Palm Phenolics
  Arms: Group B

SUMMARY:
An unpublished study by the investigators on healthy participants has shown that the supplementation of oil palm phenolics (OPP) at 250 mg is the optimum dose to demonstrate the ability to lower total and LDL cholesterol. There is no clinical evidence as yet on that optimum dosage of OPP supplementation in improving fasting lipid profile in minor hyperlipidemia subjects. The investigators hypothesize that in a clinical study, OPP supplemented to the minor hyperlipidemic participants will elicit a reduction in total and LDL cholesterol while maintaining safety and tolerability. OPP may have the potential to be positioned as natural health supplement in improving lipid profile.

DETAILED DESCRIPTION:
Oil palm phenolics (OPP) is a product filtrated from vegetation liquor of an aqueous waste stream following palm oil milling process. A novel process to recover OPP that contains a high amount of phenolic from the waste has been explored tremendously. Due to the high phenolic content, OPP has been postulated in possessing various medicinal properties such as antioxidant, anti-inflammatory, neuroprotective and anti-tumour effects.

Hyperlipidemia is a well-known risk factor for cardiovascular diseases (CVD). It can be defined as elevations of fasting total cholesterol or triglyceride concentration or both. According to a previous research, OPP supplementation to hamster animal model has shown positive effects in the reduction of total cholesterol and triglycerides as well as improvement of high-density lipoprotein cholesterol (HDL-C). In a previous study using the rabbit animal model, OPP has shown a protective effect against atherosclerosis, a condition whereby fat and cholesterol plaques are deposited inside the arteries. Based on the current evidence from the preliminary studies on OPP, the investigators hypothesize that supplementation of OPP may prevent or delay the development of CVD.

In the investigator's previous clinical trial phase I, an optimum dosage of OPP has been obtained. Therefore, the investigators proposed a phase II clinical trial to evaluate the ability of OPP to reduce the total and LDL cholesterol in minor hyperlipidemic participants.

This study will be initiated with the recruitment of 50 volunteers with minor hyperlipidemic condition. In this study, the participants will be supplemented with placebo/OPP capsules for 60 days. Participants will be required to take the placebo/OPP capsules in front of the study staff to ensure compliance. Blood samples will be withdrawn at baseline, day 30 and day 60, and will be analyzed for lipid profile, antioxidant and anti-inflammatory status. Data from this study would hopefully assist the investigator in understanding the therapeutic roles of OPP in humans under minor hyperlipidemic conditions.

ELIGIBILITY:
Inclusion Criteria:

* Elevated Fasting Total cholesterol level of more than 5.2 mmol/L
* Elevated Fasting LDL cholesterol of more than 3.36 mmol/L*
* Elevated Fasting Triglycerides of more than 1.69 mmol/L*
* Willing to remain staying in Klang Valley area in the case of Movement Control Order implementation.

Exclusion Criteria:

* Elevated Total cholesterol level of more than 6.2 mmol/L
* Elevated LDL cholesterol of more than 4.9 mmol/L
* Elevated Triglycerides of more than 5.6 mmol/L
* Smoking
* Habitual alcohol consumption
* Consuming antioxidant supplement
* Pregnant/ breastfeeding
* Medical history of cardiovascular disease, diabetes, dyslipidemia, familial hyperlipidemia, hypothyroidism, kidney disease and endocrine disease.
* Current use of lipid-lowering medication

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Changes of fasting plasma LDL cholesterol levels | Baseline, day 30, day 60 after supplementation
  This will be assessed from the Fasting Plasma LDL Cholesterol level of each participant following one month and two months supplementation.

SECONDARY OUTCOMES:
Changes of Fasting lipid profile (total cholesterol) | Baseline, day 30 and day 60 after supplementation
  This will be assessed from the Fasting Plasma Total Cholesterol level of each participant following one month and two months supplementation
Changes of Fasting lipid profile (HDL cholesterol) | Baseline,day 30 and day 60 after supplementation
  This will be assessed from the Fasting Plasma HDL Cholesterol level of each participant following one month and two months supplementation
Changes of Fasting lipid profile (Triglyceride) | Baseline,day 30 and day 60 after supplementation
  This will be assessed from the Fasting Plasma Triglyceride level of each participant following one month and two months supplementation
Changes of plasma inflammatory markers | Baseline, day 30 and day 60 after supplementation
  Inflammatory markers such as Interleukin-6, Interleukin-1beta, Tumour Necrosis Factor-alpha, Interleukin-10 and interferon-Gamma will be assessed from the plasma analysis on the fasting blood samples of each participant following one and two months of supplementation. The measurement of the plasma inflammatory markers will be performed by Multiplex assay method.
Changes of Plasma Antioxidant Levels | Baseline, day 30 and day 60 after supplementation
  Antioxidant levels such as Malonaldehyde and Superoxide dismutase will be assessed from the plasma analysis on the fasting blood samples of each participant following one and two months of supplementation. The measurement of the antioxidant levels will be performed by Using ELISA Method.
Incidence of adverse events via evaluation of renal function test | Baseline, day 30 and day 60 after supplementation
  This will be assessed by Kidney Function test from the fasting plasma analysis of each participant following one month and two months supplementation
Incidence of adverse events via evaluation of liver function test | Baseline, day 30 and day 60 after supplementation
  This will be assessed by Liver Function Test from the fasting plasma analysis of each participants following one-month and two-months supplementation
Changes of Body weight measurement | Baseline, day 30 and day 60 after supplementation
  This will be assessed by measuring the weight of each participant. Any drastic change in body weight will indicate non-compliance.

CONTACTS AND LOCATIONS:
Overall Officials: Isa Naina Mohamed, Principal Investigator — National University of Malaysia
Locations (1):
- National University of Malaysia, Cheras, WP Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fairus S, Leow SS, Mohamed IN, Tan YA, Sundram K, Sambanthamurthi R. A phase I single-blind clinical trial to evaluate the safety of oil palm phenolics (OPP) supplementation in healthy volunteers. Sci Rep. 2018 May 29;8(1):8217. doi: 10.1038/s41598-018-26384-7. PMID 29844318
- [Derived] Muhammad Ismail Tadj NB, Ibrahim NI, Tg Abu Bakar Sidik TMI, Zulfarina MS, Haji Mohd Saad Q, Leow SS, Fairus S, Naina Mohamed I. Safety and efficacy of oil palm phenolic supplementation in improving lipid profile among hyperlipidemic adults: a phase 2, randomized, double-blind, placebo-controlled clinical trial. Front Pharmacol. 2023 Jul 7;14:1190663. doi: 10.3389/fphar.2023.1190663. eCollection 2023. PMID 37484009